CLINICAL TRIAL: NCT05877690
Title: Selective Spinal Anesthesia Using Hyperbaric Prilocaine 2% Provides Better Perioperative Hemodynamic Stability for Patients With Peripheral Vascular Disease and Cardiac Dysfunction Undergoing Lower Limb Vascular Surgery
Brief Title: Selective Spinal Anaesthesia With Hyperbaric Prilocain With 2%Provides Better Perioperative Hemodynamic Stability for Patients With Peripheral Vascular Disease and Cardiac Dysfunction in Lower Limb Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zahwa Ahmed Yehya, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Selective spinal anaesthesia
Record Dates: First submitted 2023-02-23; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-03

CONDITIONS: Hemodynamic Stability
MeSH Terms: interventions — Bupivacaine; Prilocaine; Injections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Experimental)
  Interventions: Drug: Bupivacaine 0.5% Injectable Solution
- Group p (Experimental)
  Interventions: Drug: Prilocaine Hydrochloride 2% Injection

INTERVENTIONS:
Drug: Bupivacaine 0.5% Injectable Solution — Patient will be received the drug intrathecal
  Other Names: Marcaine
  Arms: Group M
Drug: Prilocaine Hydrochloride 2% Injection — Patient will be received the drug intrathecal
  Other Names: Takipril
  Arms: Group p

SUMMARY:
to compare the safety and efficacy of spinal anesthesia using Hyperbaric Prilocaine 2% versus Hyperbaric Bupivacaine 0.5% for patients with peripheral vascular disease and cardiac dysfunction.

DETAILED DESCRIPTION:
Spinal anesthesia has become increasingly popular for inpatient surgery, but, until recently, its use has been limited in ambulatory surgery due to the lack of a safe and licensed short-acting local anesthetic agent. An ideal intrathecal agent for ambulatory surgery should have a rapid onset of motor and sensory blockade, predictable regression within an acceptable time frame, and a low incidence of adverse effects. Hyperbaric Bupivacaine is a long-acting local anesthetic from the amide group and has a low incidence of transient neurological symptoms (TNS). Because of its pharmacological profile, the recovery of motor and sensory blocks is delayed compared to short-acting local anesthetics. The incidence of postoperative urinary retention with long-acting local anesthetics like bupivacaine is higher than with short-acting local anesthetics . Successful spinal anesthesia with low doses of bupivacaine between 5 and 10 mg without additives has been described for outpatients. The incidence of urinary retention was still 3.7-16%. Furthermore, with these low doses, block height becomes unpredictable, and the risk of block failure is high . Prilocaine is an amide local anesthetic with an intermediate duration of action after spinal administration. Recently, the old local anesthetics prilocaine was reintroduced in the market. It is available in the hyperbaric form and provides anesthesia for 75-90 min after spinal administration . Hyperbaric prilocaine 2% is increasingly used for spinal anesthesia in the ambulatory setting , as it has the advantage of faster recovery times than hyperbaric bupivacaine . We aimed to compare spinal anesthesia using hyperbaric prilocaine 2% and hyperbaric bupivacaine 0.5% for day case surgery in terms of sensory block, and motor block resolution times. The time for first spontaneous voiding and duration of stay in the PACU and time to home readiness.

Vascular disease and cardiac dysfunction are linked in many ways. They share common risk factors and comorbidities, and patients with systemic vascular disease often have concomitant heart disease, because the blood vessels of the heart are not spared. In patients presenting for surgery, the presence of vascular disease puts the patient at increased risk for perioperative cardiac complications, and vascular surgery poses the highest surgical risk for perioperative cardiac events.

In addition, the diseased vessels supplying critical organs depend on the perfusion pressure supplied by the heart, so any cardiac dysfunction thus amplifies the effect of poor perfusion. Patients presenting with both vascular disease and cardiac dysfunction pose a particular challenge to the anesthesiologist; although treatment goals are similar small physiologic disturbances can quickly lead to large, serious changes in clinical status.

Selective spinal anesthesia performed with a short-term hyperbaric local anesthetic could be a perfect solution, because it guarantees rapid sensory and motor block, predictable duration, and low incidence of side effects. It is usually well accepted by both patients and surgeons due to its high reliability, as it provides effective analgesia, with minimal side effects, rapid changeover times, and low costs .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of aged >18 years old. Both sexes, males and females.
* The time of surgery does not exceed 75 min.
* Compensated cardiac dysfunction
* ASA physical status: II- IV

Exclusion Criteria:

* refusal
* Allergy to the studied drugs.
* Patients with contraindications to spinal anesthesia.
* Patients with advanced decompensated cardiac, renal, hepatic disease
* Coagulopathy or thrombocytopenia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Monitoring blood pressure both systole and diastole | 75 minutes
  When, how the chang in the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ekram Abdullah, Professor, Study Chair — Assiut University
Locations (1):
- Assuit university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No